CLINICAL TRIAL: NCT02629588
Title: Effectiveness of Sensory Stimulation for Person in a Coma or Persistent Vegetative State After Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Rene L. Padilla, Associate Professor of Occupational Therapy, Creighton University
Other Study IDs: AJOT/2015/021022
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Brain Injuries
Keywords: Coma; Persistent Vegetative State; Sensory Stimulation
MeSH Terms: conditions — Brain Injuries; Coma; Persistent Vegetative State

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Persons in coma or vegetative state: People who survived TBI have a period of complete unconsciousness or coma with no awareness of themselves or their surroundings received multimodal or unimodal sensory stimulation.People in a coma are unaware and unresponsive, but not asleep as there is no sleep-wake cycle. While in a coma, people are unable to speak, follow commands or open their eyes. The person in coma may have a simple reflex in response to touch or pain, but essentially there is no meaningful response to external stimuli. There is an absence of awareness of self and the environment, even under conditions of vigorous external stimulation. Coma can last from hours to days, depending on the severity of the brain damage, and sometimes a person can remain in a comatose state for months and even years.
  Interventions: Behavioral: Multimodal or Unimodal Sensory stimulation

INTERVENTIONS:
Behavioral: Multimodal or Unimodal Sensory stimulation — multimodal sensory stimulation, unimodal sensory stimulation, auditory stimulation, complex stimulation, median nerve stimulation.

SUMMARY:
Appraised the empirical evidence of effectiveness of sensory stimulation to improve arousal and alertness for persons in a coma or persistent vegetative state after traumatic brain injury (TBI). Databases were searched and nine articles met inclusion criteria.

DETAILED DESCRIPTION:
Background: Traumatic brain injury (TBI) accounts for approximately 50,000 deaths in the United States each year. About 17% of survivors have a period of "coma". Duration of coma contributes significantly to functional outcomes.

Objective: To appraise the evidence of effectiveness of sensory stimulation to improve arousal and alertness for persons in a coma or persistent vegetative state after TBI.

Data Sources and Study Eligibility Criteria: Databases searched included Medline, PsycINFO, CINAHL, OTseeker, and the Cochrane Database of Systematic Reviews. The search was limited to outcomes studies in the hierarchy described by Sackett and colleagues (1996), published in English in peer-reviewed journals between 2006 and 2014.

ELIGIBILITY:
Inclusion Criteria:

* in coma or persistent vegetative state after traumatic brain injury

Exclusion Criteria:

* coma or persistent vegetative state not caused by traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons in a coma or persistent vegetative state (Glasgow Coma Scale below 8) after traumatic brain injury
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Glasgow Coma Scale | 0-30 days post injury

CONTACTS AND LOCATIONS:
Overall Officials: Rene L Padilla, PhD, Principal Investigator — Creighton University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbate C, Trimarchi PD, Basile I, Mazzucchi A, Devalle G. Sensory stimulation for patients with disorders of consciousness: from stimulation to rehabilitation. Front Hum Neurosci. 2014 Aug 11;8:616. doi: 10.3389/fnhum.2014.00616. eCollection 2014. No abstract available. PMID 25157226
- [Background] Alali AS, Fowler RA, Mainprize TG, Scales DC, Kiss A, de Mestral C, Ray JG, Nathens AB. Intracranial pressure monitoring in severe traumatic brain injury: results from the American College of Surgeons Trauma Quality Improvement Program. J Neurotrauma. 2013 Oct 15;30(20):1737-46. doi: 10.1089/neu.2012.2802. Epub 2013 Jul 11. PMID 23731257
- [Background] Li N, Yang Y, Glover DP, Zhang J, Saraswati M, Robertson C, Pelled G. Evidence for impaired plasticity after traumatic brain injury in the developing brain. J Neurotrauma. 2014 Feb 15;31(4):395-403. doi: 10.1089/neu.2013.3059. Epub 2013 Dec 10. PMID 24050267
- [Background] Wood RL, Winkowski TB, Miller JL, Tierney L, Goldman L. Evaluating sensory regulation as a method to improve awareness in patients with altered states of consciousness: a pilot study. Brain Inj. 1992 Sep-Oct;6(5):411-8. doi: 10.3109/02699059209008137. PMID 1393174
- [Background] Becker JM, Shanley PJ. Defending the healthcare fraud case: parallel proceedings and collateral consequences. Del Med J. 1992 Jun;64(6):393-8. No abstract available. PMID 1451851
- [Background] Cremer OL, van Dijk GW, van Wensen E, Brekelmans GJ, Moons KG, Leenen LP, Kalkman CJ. Effect of intracranial pressure monitoring and targeted intensive care on functional outcome after severe head injury. Crit Care Med. 2005 Oct;33(10):2207-13. doi: 10.1097/01.ccm.0000181300.99078.b5. PMID 16215372
- [Background] Duff D. Review article: altered states of consciousness, theories of recovery, and assessment following a severe traumatic brain injury. Axone. 2001 Sep;23(1):18-23. PMID 14621499
- [Background] Dunn W. The sensations of everyday life: empirical, theoretical, and pragmatic considerations. Am J Occup Ther. 2001 Nov-Dec;55(6):608-20. doi: 10.5014/ajot.55.6.608. PMID 12959225
- [Background] Giacino JT, Whyte J, Bagiella E, Kalmar K, Childs N, Khademi A, Eifert B, Long D, Katz DI, Cho S, Yablon SA, Luther M, Hammond FM, Nordenbo A, Novak P, Mercer W, Maurer-Karattup P, Sherer M. Placebo-controlled trial of amantadine for severe traumatic brain injury. N Engl J Med. 2012 Mar 1;366(9):819-26. doi: 10.1056/NEJMoa1102609. PMID 22375973
- [Background] Hendricks HT, Geurts AC, van Ginneken BC, Heeren AJ, Vos PE. Brain injury severity and autonomic dysregulation accurately predict heterotopic ossification in patients with traumatic brain injury. Clin Rehabil. 2007 Jun;21(6):545-53. doi: 10.1177/0269215507075260. PMID 17613585
- [Background] Lannin NA, Cusick A, McLachlan R, Allaous J. Observed recovery sequence in neurobehavioral function after severe traumatic brain injury. Am J Occup Ther. 2013 Sep-Oct;67(5):543-9. doi: 10.5014/ajot.2013.008094. PMID 23968792
- [Background] Sackett DL, Rosenberg WM, Gray JA, Haynes RB, Richardson WS. Evidence based medicine: what it is and what it isn't. 1996. Clin Orthop Relat Res. 2007 Feb;455:3-5. No abstract available. PMID 17340682
- [Result] Abbasi M, Mohammadi E, Sheaykh Rezayi A. Effect of a regular family visiting program as an affective, auditory, and tactile stimulation on the consciousness level of comatose patients with a head injury. Jpn J Nurs Sci. 2009 Jun;6(1):21-6. doi: 10.1111/j.1742-7924.2009.00117.x. PMID 19566636
- [Result] Cheng L, Gosseries O, Ying L, Hu X, Yu D, Gao H, He M, Schnakers C, Laureys S, Di H. Assessment of localisation to auditory stimulation in post-comatose states: use the patient's own name. BMC Neurol. 2013 Mar 18;13:27. doi: 10.1186/1471-2377-13-27. PMID 23506054
- [Result] DeFina PA, Fellus J, Thompson JW, Eller M, Moser RS, Frisina PG, Schatz P, Deluca J, Zigarelli-McNish M, Prestigiacomo CJ. Improving outcomes of severe disorders of consciousness. Restor Neurol Neurosci. 2010;28(6):769-80. doi: 10.3233/RNN-2010-0548. PMID 21209492
- [Result] Di Stefano C, Cortesi A, Masotti S, Simoncini L, Piperno R. Increased behavioural responsiveness with complex stimulation in VS and MCS: preliminary results. Brain Inj. 2012;26(10):1250-6. doi: 10.3109/02699052.2012.667588. Epub 2012 May 22. PMID 22616735
- [Result] Megha M, Harpreet S, Nayeem Z. Effect of frequency of multimodal coma stimulation on the consciousness levels of traumatic brain injury comatose patients. Brain Inj. 2013;27(5):570-7. doi: 10.3109/02699052.2013.767937. Epub 2013 Mar 8. PMID 23473238
- [Result] Meyer MJ, Megyesi J, Meythaler J, Murie-Fernandez M, Aubut JA, Foley N, Salter K, Bayley M, Marshall S, Teasell R. Acute management of acquired brain injury Part III: an evidence-based review of interventions used to promote arousal from coma. Brain Inj. 2010;24(5):722-9. doi: 10.3109/02699051003692134. PMID 20334468
- [Result] Noe E, Olaya J, Navarro MD, Noguera P, Colomer C, Garcia-Panach J, Rivero S, Moliner B, Ferri J. Behavioral recovery in disorders of consciousness: a prospective study with the Spanish version of the Coma Recovery Scale-Revised. Arch Phys Med Rehabil. 2012 Mar;93(3):428-33.e12. doi: 10.1016/j.apmr.2011.08.048. Epub 2012 Jan 24. PMID 22277244
- [Result] Oh H, Seo W. Sensory stimulation programme to improve recovery in comatose patients. J Clin Nurs. 2003 May;12(3):394-404. doi: 10.1046/j.1365-2702.2003.00750.x. PMID 12709114
- [Derived] Padilla R, Domina A. Effectiveness of Sensory Stimulation to Improve Arousal and Alertness of People in a Coma or Persistent Vegetative State After Traumatic Brain Injury: A Systematic Review. Am J Occup Ther. 2016 May-Jun;70(3):7003180030p1-8. doi: 10.5014/ajot.2016.021022. PMID 27089287
- See also: Agency for Healthcare Research and Quality, U.S. Preventive Task Force. (2012). Grade definitions. — http://www.uspreventiveservicestaskforce.org/Page/Name/grade-definitions